CLINICAL TRIAL: NCT06958614
Title: Efficacy and Safety of Primary Prophylactic Pegylated Recombinant Human Granulocyte Colony-Stimulating Factor During Definitive Concurrent Chemoradiotherapy for Inoperable Stage II-III Non-Small Cell Lung Cancer: A Prospective Cohort Study
Brief Title: Prophylactic PEG-rhG-CSF During cCRT in LA-NSCLC
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIANYANG WANG, Professor,MD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: 19/216-2000
Record Dates: First submitted 2025-03-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Stage II-III Non-small Cell Lung Cancer; Concurrent Chemotherapy; Conditions Influencing Health Status
Keywords: Pegylated recombinant human granulocyte colony-stimulating factor; Non-small cell lung cancer; concurrent chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Primary Prophylactic Pegylated Recombinant Human Granulocyte Colony-Stimulating Factor — The experimental group received prophylactic PEG-rhG-CSF 48 hours after chemotherapy

SUMMARY:
Objective: To evaluate the efficacy and safety of prophylactic use of pegylated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF) during definitive concurrent chemoradiotherapy (cCRT) in patients with inoperable stage II-III non-small cell lung cancer (NSCLC).

Methods: A prospective observational cohort study was conducted on patients receiving definitive cCRT. The radiation therapy technique uses intensity modulated radiation therapy (IMRT) and involves field irradiation. It protects more normal tissue from exposure.Chemotherapy regimens included platinum-based doublet combinations: etoposide plus cisplatin (every 28 days), pemetrexed plus platinum (every 21 days), or paclitaxel plus platinum (weekly, only for control group) .

Patients were followed up at one month post-treatment, then every three months for the two year, and every six months thereafter until disease progression.

In the study group, patients received subcutaneous injections of PEG-rhG-CSF (6 mg for patients weighing ≥45 kg, 3 mg for patients <45 kg) 48 hours after each chemotherapy cycle during cCRT. In the control group, patients received guideline-based supportive treatment. Radiotherapy was halted or chemotherapy was delayed when grade 3 or more (G3+) toxicities happened.

Endpoints:Primary endpoint was incidence of G3+ neutropenia during radiotherapy and one month post-radiotherapy. Complete blood counts were monitored weekly during cCRT and for one month post-treatment or as deemed necessary by the physician.

Following the completion of cCRT and the resolution of acute side effects, patients were followed up at one month post-treatment, then every three months for the first year, and every six months thereafter until disease progression.

Statistical Analysis:The inverse probability of treatment weighting (IPTW) algorithm was applied to balance differences between groups in terms of age, gender, smoking, clinical stage, KPS score, induction therapy received or not, ensuring the reliability of the study results. Statistical analysis was performed using R software (version 4.4.1). All tests were two-sided, with a P-value <0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis

   * Histologically confirmed stage II-III non-small cell lung cancer (NSCLC)
2. Treatment Plan

   * Planned to receive concurrent platinum-based chemotherapy with radiotherapy (cCRT)
3. Demographics

   * Age 18-80 years
4. Performance Status

   * Karnofsky Performance Status (KPS) ≥70
5. Organ Function

   * Renal function: Creatinine clearance ≥60 mL/min
   * Hepatic function: Total bilirubin ≤1.5×ULN, AST/ALT ≤2.5×ULN
   * Absolute neutrophil count ≥2.0×10⁹/L
   * Platelets ≥100×10⁹/L
   * Hemoglobin ≥10 g/dL

Exclusion Criteria:

1. Active Malignancies

   * Concurrent diagnosis of active malignancies (excluding: non-melanoma skin cancer, carcinoma in situ, or malignancies in complete remission for ≥5 years)
2. Infectious/Immunological Conditions

   * Active systemic infection requiring intravenous antimicrobial therapy
   * Uncontrolled autoimmune diseases (defined as requiring systemic immunosuppressants at doses >10 mg/day prednisone equivalent within 30 days prior to screening)
3. Hypersensitivity Reactions

   * Allergy to PEG-rhG-CSF or other biological products derived from genetically engineered Escherichia coli
4. Neuropsychiatric Impairments

   * Severe psychiatric disorders (e.g., schizophrenia, major depressive disorder with suicidal ideation) requiring hospitalization within 6 months)
5. Prior Radiotherapy

   * History of thoracic radiotherapy involving >30% lung parenchyma or mean heart dose >20 Gy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Definitive Concurrent Chemoradiotherapy for Inoperable Stage II-III Non-Small Cell Lung Cancer，Patients received prophylactic PEG-rhG-CSF 48 hours after chemotherapy.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Grade 3 or more (G3+) neutropenia | From the first day of radiotherapy to one month after the end of radiotherapy
  According to the Radiation Therapy Oncology Group (RTOG) acute radiation injury grading scale

SECONDARY OUTCOMES:
treatment delays | Chemotherapy delay was defined as a delay of ≥7 days
  Chemotherapy delay
interruptions | Break in radiotherapy of ≥3 days
  Radiotherapy interruption
G3+ thrombocytopenia and anemia | From the first day of radiotherapy to one month after the end of radiotherapy
  According to the Radiation Therapy Oncology Group (RTOG) acute radiation injury grading scale
G2+ acute radiation esophagitis (RE) and pneumonitis (RP) | From the first day of radiotherapy to six month after the end of radiotherapy
  According to the Radiation Therapy Oncology Group (RTOG) acute radiation injury grading scale
progression-free survival (PFS) | assessed up to 72 months
  the time from the start of cCRT to the first event of disease progression
overall survival (OS) | assessed up to 72 months
  the time from the start of cCRT to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

DOCUMENTS (1):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT06958614/Prot_000.pdf